CLINICAL TRIAL: NCT06887101
Title: Impact of Stress on Cardiovascular Events in Patients with Peripheral Arterial Disease
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Essen (Other)
Collaborators: Universität Duisburg-Essen (Other)
Responsible Party: Sponsor
Other Study IDs: 23-11092-BO
Record Dates: First submitted 2025-02-27; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-01

CONDITIONS: Peripheral Arterial Disease
Keywords: vascular diseases; cardiovascular diseases; ischemia; arteriosclerosis; stress
MeSH Terms: conditions — Peripheral Arterial Disease; Vascular Diseases; Cardiovascular Diseases; Ischemia; Arteriosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Hair cortisol. Standard blood tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with peripheral arterial disease.: No control group is planned for this trial.

SUMMARY:
Atherosclerotic cardiovascular disease is the leading cause of morbidity and mortality worldwide. Patients with peripheral arterial disease are at increased risk suffering from major adverse cardiac and limb events. Acute and chronic stress affect the cardiovascular system. Long-term negative stressors lead to cardiovascular diseases and can aggravate already existing cardiovascular diseases. However, current guidelines on cardiovascular disease prevention highlight stress as a cardiovascular risk factor there is a lack of consensus about the definition and measurement of stress. The aim of the proposed trial is to evaluate different stress measuring methods in patients with PAD depending on the occurrence of cardiovascular events.

DETAILED DESCRIPTION:
Based on World Health Organization data, atherosclerotic cardiovascular disease (CVD) is the leading cause of morbidity and mortality worldwide. Peripheral arterial disease (PAD) is a poly-vascular disease in multiple arterial beds mostly associated with high atherosclerotic burden. It is estimated that around 50 million people in Europe alone suffer from PAD and the prevalence increases with age. The cause of CVD, such as PAD, coronary artery disease (CAD) or cerebrovascular disease, is atherosclerosis, a systemic chronic inflammatory vascular disease. Patients with CVD are at increased risk of life-threatening complications such as acute limb events, stroke and myocardial infarction combined with an impaired quality of life.

Acute and chronic stress affect the cardiovascular system. Numerous studies have shown the relationship between chronic stress and cardiovascular diseases. On the one hand, permanent negative stressors lead to cardiovascular diseases via different pathways such as the hypothalamic-pituitary-adrenal (HPA) axis or the autonomic nervous system, and, on the other hand, stress can aggravate an already existing CVD. In addition, cardiovascular risk factors like hypertension and hypercholesteremia are negatively influenced by stress. Stress as a cardiovascular risk factor is receiving increasing attention, leading to its recognition in current guidelines on cardiovascular disease prevention.

Due to the demographic development of an ageing population and the simultaneous increase in atherogenic risk factors, a further rise of patients with CVD will be expected in the future. Thus, sufficient assessment of cardiovascular risk in patients with PAD and adequate stress evaluation are elementary. However, there is a lack of consensus about the definition and measurement of stress.

Therefore, the investigators aim to evaluate and compare the efficiency of different stress measuring methods depending on the occurrence of major adverse cardiovascular events (MACE) and major adverse limb events (MALE) in patients with PAD.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of lower extremity PAD based on:

* Limb bypass surgery or
* aorta-femoral bypass surgery or
* percutaneous transluminal angioplasty revascularization of the iliac or infrainguinal arteries or
* limb or foot amputation for arterial vascular disease or
* intermittent claudication and one or more of either an ankle brachial index (ABI) of less than 0.90 or a peripheral artery stenosis (≥50%) documented by angiography or duplex ultrasound or carotid revascularization or asymptomatic carotid artery stenosis of at least 50% diagnosed by duplex ultrasound or angiography

Exclusion Criteria:

* atrial fibrillation
* high premature ventricular contractions burden
* pacemaker with constant ventricular pacing
* antiarrhythmic drugs class I or III

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The recruitment process and examinations will take place at the Department of Cardiology and Vascular Medicine, West German Heart and Vascular Center, University Hospital Essen.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Myocardial Infarction (MI), Ischemic Stroke, Acute Limb Ischemia (ALI), Coronary Heart Disease (CHD) Death, or chronic limb ischemia and amputation | Baseline, after 6 months, after 12 months
  Based on the COMPASS trial MACE and MALE includes the composite of cardiovascular death, myocardial infarction, acute limb ischaemia, chronic limb ischaemia and amputation. MACE and MALE will be evaluated at baseline and after 6 and 12 months
Pychological stress | Baseline, after 6 months, after 12 months
  Pychological stress is evaluated by a composite psychometric measure of stress level by using a mean rank at baseline and after 1 year. It is based on a published RCT by Blumenthal et al. and includes the Beck Depression Inventory II (BDI-II), State-Trait Anxiety inventory (STAI), Patient-Reported Outcomes Measurement Information System (PROMIS) Anger, General Health Questionnaire (GHQ) and Perceived Stress Scale (PSS). A range from 1 to 147 was present with higher scores suggestive of better function
Heart rate variability (HRV) | Baseline, after 6 months, after 12 months
  Heart rate variability (HRV) is an indirect marker of autonomic nervous system activity and describes the oscillations between the R-R intervals in the electrocardiogram. It allows a relatively superficial insight into the heart-brain interaction and reflects the psycho-emotional status such as stress or anxiety. According to the guidelines we chose a short-time HRV with 5 minutes of recording
Proinflammatory mediators - IL-6 | Baseline, after 6 months, after 12 months
  IL-6 is measured in pg/ml. Standard value is under 2.7 pg/ml. Higher values indicate an increased stress level
Proinflammatory mediators - IL-1ß | Baseline, after 6 months, after 12 months
  IL-1ß is measured in pg/ml. Standard value is under 5 pg/ml. Higher values indicate an increased stress level
Proinflammatory mediators - TNFalpha | Baseline, after 6 months, after 12 months
  TNFalpha is measured in pg/ml. Standard value is under 2.8 pg/ml. Higher values indicate an increased stress level
Proinflammatory mediators - hsCRP | Baseline, after 6 months, after 12 months
  High sensitive-c-reactive protein (hsCRP) is measured in mg/dl. Standard value is under 0.02 mg/dl. Higher values indicate an increased stress level
Hair cortisol concentration | Baseline, after 6 months, after 12 months
  Hair cortisol is reliable biomarker of chronic stress that offers a retrospective non-invasive measurement of long-term HPA-axis activity over several weeks or months. The cortisol concentration, measured in pg/ml, of a 3 cm hair segment using liquid chromatography tandem mass spectrometry will be analyzed. Higher values indicate an increased stress level

SECONDARY OUTCOMES:
Health-related quality of life | Baseline, after 6 months, after 12 months
  We will apply two instrument to measure health-related quality of life. Namely the Short Form-36 health questionnaire and the European Quality of Life 5 Dimensions 5 Level survey (EQ-5D-5L). The SF-36 is an eight-dimensional scale consisting of 36 items. It assesses health-related quality of life based on physical, social, and psychological functioning, role behavior due to physical and psychological functional impairment, physical pain, general health perception, and vitality. The EQ-5D-5L consists of five health-related dimensions that can be assessed at five levels. In addition, the questionnaire contains a visual analog scale for assessing general health
Ankle-brachial index (ABI) | Baseline, after 6 months, after 12 months
  The lower systolic ankle pressure is set in relation to the systolic blood pressure of the upper extremity. The lowest calculated ABI will be used. Normal values are 0.9 to 1.2. ABI values below 0.9 are indicative of PAD, with an ABI below 0.5 showing severe limb ischaemia
Changes in functional capacity | Baseline, after 6 months, after 12 months
  Changes in functional capacity will be recorded using the established 6-minute walk test
LDL-Cholesterol | Baseline, after 6 months, after 12 months
  Low density lipoprotein (LDL) is measured in mg/dl
Serum-cortisol | Baseline, after 6 months, after 12 months
  Serum-Cortisol is measured in mol/l
Depression symptoms (BDI-II) | Baseline, after 6 months, after 12 months
  The BDI-II is a self-report questionnaire comprising 21 items that assess depression severity. Its reliability and validity have been established through various studies among diverse populations and cultural backgrounds. Higher scores indicates increased depression symptoms
Anxiety symptoms (STAI) | Baseline, after 6 months, after 12 months
  The STAI is the most authoritative tool for assessing anxiety in adults, precisely distinguishing between transient "state anxiety" and persistent "trait anxiety". The STAI measures anxiety with 20 items and has a range of 20 to 80. A higher score indicates more pronounced anxiety.
PROMIS-Anger Scale | Baseline, after 6 months, after 12 months
  The PROMIS Anger scale comprises eight items that evaluate various aspects of anger. Scores on the scale range from 8 to 40, with higher scores indicating greater levels of anger
GHQ | Baseline, after 6 months, after 12 months
  The GHQ assesses general distress and consists of 12 items. Respondents' scores range from 0 to 36, where higher scores correspond to increased distress
Perceived Stress Scale | Baseline, after 6 months, after 12 months
  The Perceived Stress Scale-10 item version is a short tool for the assessment of how individuals perceive stress in their lives. The values range from 0 to 40. Higher values indicate higher perceived stress.
  (l) In-treatment assessments: at the start of each intervention module (weekly), the following assessment instruments will be applied: Distress Thermometer (DT), Patient Health Questionnaire-4 (PHQ-4) and self-generated measures to assess coping skills and self-efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology and Vascular Medicine, West German Heart and Vascular Center, University Hospital Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: after publication
Access Criteria: contact PI